CLINICAL TRIAL: NCT00108771
Title: Double-Blind, Parallel, Randomized, Placebo-Controlled 12-Week Efficacy and Safety Assessment of ZR-02-01 in the Treatment of Chronic, Moderate to Severe Osteoarthritis (OA) Pain
Brief Title: Fentanyl Transdermal Matrix Patch ZR-02-01 to Treat Chronic, Moderate to Severe Osteoarthritis (OA) Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZMF-202
Record Dates: First submitted 2005-04-18; First posted 2005-04-19 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Pain
Keywords: Pain; Chronic Pain; Osteoarthritis Pain; Osteoarthritis
MeSH Terms: conditions — Pain; Chronic Pain; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZR-02-01 matrix fentanyl Patch (Experimental): ZR-02-01 matrix fentanyl patch
  Interventions: Drug: ZR-02-01 Fentanyl Transdermal Matrix Patch
- Placebo Patch (Placebo Comparator)
  Interventions: Drug: Placebo Patch

INTERVENTIONS:
Drug: ZR-02-01 Fentanyl Transdermal Matrix Patch — Study patches were replaced every 72 hours and were to be applied on the upper chest or lateral aspect of the upper arms. The patch application sites were to be rotated so the patch was not applied to the same skin site for successive applications. Patients were supplied with Tegaderm if needed to keep the patches adhered during the 72 hour wear period.
  Other Names: ZR-02-01
  Arms: ZR-02-01 matrix fentanyl Patch
Drug: Placebo Patch — Study patches were replaced every 72 hours and were to be applied on the upper chest or lateral aspect of the upper arms. The patch application sites were to be rotated so the patch was not applied to the same skin site for successive applications. Patients were supplied with Tegaderm if needed to keep the patches adhered during the 72 hour wear period
  Other Names: Placebo Transdermal Matrix Patch
  Arms: Placebo Patch

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the Matrix Fentanyl Patch ZR-02-01 in providing pain relief.

DETAILED DESCRIPTION:
This study will evaluate the analgesic efficacy of the matrix fentanyl patch. The study will be conducted in non-opioid tolerant patients with moderate to severe osteoarthritis (OA) pain. This patient population was chosen in anticipation that the patients are otherwise healthy adults being treated with NSAIDs (Nonsteroidal Anti-inflammatory Drugs) or acetaminophen or who have received intermittent opioid analgesic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 40 and 75 years of age suffering from moderate to severe chronic pain caused by osteoarthritis.

Exclusion Criteria:

* Patient is already taking chronic opioids or has a history of substance abuse or has a substance abuse disorder.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2004-04; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
WOMAC Knee and Hip Osteoarthritis Index | 12 weeks
  The Pain,Stiffness and Physical Function subscales of the WOMAC Knee and Hip Osteoarthritis Index (5-point Likert scale: none through extreme) was employed. The subscales consist of 24 questions (5 pain, 2 stiffness and 17 physical function)

SECONDARY OUTCOMES:
Number of participants with adverse events | 12 weeks
TOPS survey | 12 weeks
  To document outcomes following pain therapy with ZR-02-01 using the TOPS survey, a disease-specific measure of health

CONTACTS AND LOCATIONS:
Overall Officials: Frank Farmer, Jr, MD, Principal Investigator — Radiant Research
Locations (13):
- United States (13):
  - Arizona Reserach Center, Phoenix, Arizona
  - Redpoint Research, Phoenix, Arizona
  - Sharp Rees-Stealy Medical Group, San Diego, California
  - San Diego Arthritis Medical Clinic, San Diego, California
  - Boling Clinical Trials, Upland, California
  - Radiant Research, Daytona Beach, Florida
  - Ocala Rheumatology, Ocala, Florida
  - Tampa Medical Group, Tampa, Florida
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - Pain Trials Center - Brigham & Women's Hospital, Boston, Massachusetts
  - Phase III Clinical Trials, Fall River, Massachusetts
  - Beth Israel Medical Center, New York, New York
  - Analgesic Development Ltd., New York, New York